CLINICAL TRIAL: NCT04021056
Title: Observational Study on Patients With Hepatocellular Carcinoma (HCC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Jinlin Hou, Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFHCC-01
Record Dates: First submitted 2019-04-23; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
This is an ongoing, longitudinal, single centre, observational, retro-prospective clinical cohort study of patients with HCC in usual clinical practice. All the HCC patients diagnosed and treated in Liver Cancer Center, Nanfang Hospital are consecutively collected and followed up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HCC;
* Age ≥ 16 years;
* Received treatment targeting for HCC at least once, including operation, ablation, TACE, sorafenib, radiotherapy, chemotherapy, etc;
* Good compliance with clinical treatment.

Exclusion Criteria:

* Diagnosed as other pathological types such as cholangiocarcinoma, or mixed liver cancer;
* Received only traditional Chinese medicine or symptomatic supportive treatment; (3) survival time ≤ 7 days;
* HCC diagnosed after liver transplantation;
* Poor compliance or important data deficient.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed and treated as HCC in Liver Cancer Center, Nanfang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the overall survival rate of all HCC patients | 10 years
  In order to identify the potential influence factors of HCC patients survival
Evaluate the recurrence free survival rate of HCC patients after curative treatments | 10 years
  In order to identify the potential influence factors of tumor recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China